CLINICAL TRIAL: NCT06683131
Title: IMpact of PCSK9 inhibitoR initiatiOn Before Percutaneous Coronary Intervention on Coronary microVascular Dysfunction and Events for Acute Myocardial Infarction: a Multi-center, Open-label, Randomized, Controlled Trial
Brief Title: Effectiveness of Proprotein Convertase Subtilisin/Kexin Type 9 (PCSK9) Inhibitor Initiation Before Percutaneous Coronary Intervention on Acute Myocardial Infarction Patients
Acronym: IMPROVE-AMI
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: The Affiliated Hospital of Xuzhou Medical University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: XYFY2024-KL537-01
Record Dates: First submitted 2024-11-08; First posted 2024-11-12 (Actual); Last update posted 2025-11-21 (Actual); Status verified 2024-11

CONDITIONS: Acute Myocardial Infarction (AMI)
Keywords: Acute Myocardial Infarction; tafolecimab; PCSK9; Coronary Microvascular Dysfunction; Major adverse cardiovascular events; monoclonal antibody against proprotein convertase subtilisin/kexin type 9; LDL-C

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- PCSK9 inhibitor (PCSK9i) group (Experimental): Participants receive PCSK9i tafolecimab and standard of care (SoC) of acute myocardial infarction
  Interventions: Drug: Tafolecimab
- Control group (No Intervention): Participants receive SoC of acute myocardial infarction

INTERVENTIONS:
Drug: Tafolecimab — 450mg of tafolecimab (150mg each one) was injected subcutaneously before primary PCI and then 150mg subcutaneously injected every half a month till totally 12 months.
  Arms: PCSK9 inhibitor (PCSK9i) group

SUMMARY:
The goal of this clinical trial is to learn if drug tafolecimab works to treat participants with acute myocardial infarction (AMI) scheduled for primary percutaneous coronary intervention (PCI). It will also learn about the safety of drug tafolecimab. The main questions it aims to answer are:

* Does drug tafolecimab lower the risk of 1-year major adverse cardiovascular events?
* Does drug tafolecimab improve the coronary microvascular dysfunction?
* What medical problems do participants have when administering drug tafolecimab by injection? Researchers will compare the results administering drug tafolecimab or not to see if drug tafolecimab works to treat AMI.

Participants will:

* Administer drug tafolecimab by injection or not every month for 12 months
* Receive the standard of care of AMI
* Complete the measurement of coronary angiography-derived microcirculation resistance index after PCI
* Complete cardiac magnetic resonance after PCI if available
* Visit the clinic at 1,6,12 months after the first administration for checkups and tests
* Report any discomfort, event or queries at any time

ELIGIBILITY:
Inclusion Criteria:

* Adults 18-75 years old
* AMI diagnosed according to the latest guidelines, including ST-segment elevation myocardial infarction (STEMI) and non-ST-segment elevation myocardial infarction (NSTEMI)

  * The requirement for STEMI was that primary PCI was scheduled within 12 hours of onset.
  * The requirement for NSTEMI was that coronary angiography was scheduled within 2 hours for very high-risk participants and within 24 hours for high-risk participants .
* Regardless of baseline LDL-C levels
* Participants voluntarily took part in this study and signed informed consent

Exclusion Criteria:

* Previous or ongoing treatment for any PCSK9i
* Allergy to PCSK9i, statins, or any of the drug ingredients used during the trial
* History of hemorrhagic cerebrovascular disease
* History of old myocardial infarction/chronic heart failure
* History of PCI or coronary artery bypass grafting (CABG) or preparation for CABG
* Above Killip level II
* Prolonged cardiopulmonary resuscitation (>20min)
* Definite mechanical complications (including perforation of the interventricular septum, or rupture of the papillary tendon bundle or the left ventricular free wall)
* malignant arrhythmia
* Severe uncontrolled infection, bleeding disorder, end-stage renal disease, severe liver disease, endocrine dysfunction, or the expected less than 1 year survival of malignant tumors
* Pregnant or lactating women
* Participate in other clinical trials

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1160 (Estimated)
Dates: Start 2025-11-20 (Estimated); Primary Completion 2027-11-30 (Estimated); Study Completion 2027-11-30 (Estimated)

PRIMARY OUTCOMES:
Rate of major adverse cardiovascular events (MACEs) | From enrollment to 1 year after primary percutaneous coronary intervention
  MACEs including cardiovascular death, nonfatal myocardial infarction, unplanned ischemia-driven revascularization, nonfatal stroke, hospitalization for heart failure

SECONDARY OUTCOMES:
Number of participants with coronary microvascular dysfunction (CMD) | Immediately after primary percutaneous coronary intervention
  Measurement of coronary angiography-derived microcirculation resistance index (caIMR)
Number of participants with coronary microvascular dysfunction (CMD) | 3-7 days after primary percutaneous coronary intervention
  Infarct size (IS), intramyocardial hemorrhage (IMH) and microvascular obstruction (MVO) assessed by cardiac magnetic resonance
Concentration of low density lipoprotein cholesterol (LDL-C) | Both 1 month and 1 year after primary percutaneous coronary intervention
  The measurement of LDL-C level and number of participants reaching the target according to current guidelines
Rate of malignant arrhythmia | 1 month after primary percutaneous coronary intervention
  These include sudden cardiac death (SCD), sudden death survival (aborted SCD), appropriate implantable cardioverter defibrillator (ICD) interventions, and persistent ventricular arrhythmias monitored by a 72-hour holter electrocardiogram.

CONTACTS AND LOCATIONS:
Overall Officials: Yong Huo, M.D. and Ph.D., Study Chair — Peking University First Hospital; Yuan Lu, M.D. and Ph.D., Principal Investigator — The Affiliated Hospital of Xuzhou Medical University
Locations (13):
- China (13):
  - Taihe County People's Hospital, Fuyang, Anhui
  - The Fifth People's Hospital of Huai'an City, Huai'an, Jiangsu
  - Lianyungang Municipal Dongfang Hospital, Lianyungang, Jiangsu
  - Jiangsu Provincial Hospital of Traditional Chinese Medicine, Nanjing, Jiangsu
  - Jiangsu Provincial People's Hospital (The First Affiliated Hospital of Nanjing Medical University), Nanjing, Jiangsu
  - The Fourth Affiliated Hospital of Nanjing Medical University, Nanjing, Jiangsu
  - Suqian Hospital of Jiangsu Provincial People's Hospital, Suqian, Jiangsu
  - The affiliated hospital of Xuzhou Medical University, Xuzhou, Jiangsu
  - Suining County People's Hospital, Xuzhou, Jiangsu
  - Xuzhou Central Hospital, Xuzhou, Jiangsu
  - Xuzhou Mining Group General Hospital, Xuzhou, Jiangsu
  - Peking University First Hospital, Beijing
  - Shanghai Tenth People's Hospital, Shanghai

IPD SHARING:
Plan to Share IPD: No
Participants do not consent to the data sharing about themselves. IPD involves privacy and ethical issues.